CLINICAL TRIAL: NCT04061850
Title: Ibrutinib for Relapsed or Refractory Mantle Cell Lymphoma: Multicenter Retrospective Analysis
Brief Title: Ibrutinib for Relapsed or Refractory Mantle Cell Lymphoma
Acronym: MCLRR
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, MD, Ph.D, Professor of Hematology-Oncology, Samsung Medical Center
Other Study IDs: SMC 2019-04-142
Record Dates: First submitted 2019-08-14; First posted 2019-08-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To review the efficacy and the safety of ibrutinib in patients with relapsed or refractory mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
# Background and Rationale Mantle cell lymphoma (MCL) is a rare subtype of lymphoma, accounting for about 3-6% of all non-Hodgkin's lymphoma. It is clinically prevalent in the elderly and men, commonly with gastrointestinal tract involvement. Since about 80% of patients present with advanced stage disease at diagnosis, the prognosis is very poor. Mantle cell lymphoma is less frequent in Korean than in Western countries, accounting for about 2% of all non-Hodgkin's lymphoma cases, with very poor treatment outcome as Western countries.

In Korea, the clinical information about patients with MCL is very scarce so far and does not reflect recent treatment patterns. Firstly, the incidence in Korea is relatively lower than that in Western countries, with only about 100 patients a year. Secondly, due to substandard national health insurance regulations in Korea, it was not until recently that ibrutinib for relapsed/refractory MCL was approved for coverage by the National Health Insurance. In this context, the study was designed to investigate the efficacy and safety of ibrutinib in patients with relapsed or refractory MCL in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MCL diagnosed by a pathologist (based on the WHO 2017 classification)

  1. mantle cell lymphoma
  2. leukemic nonnodal mantle cell lymphoma
  3. in situ mantle cell neoplasia
* Aged ≥ 19 years
* Relapsed or refractory patients treated with ibrutinib, including relapse after autologous stem cell transplantation

Exclusion Criteria:

* Patients whose clinical and pathological data are not available
* Patients who were not treated with ibrutinib

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Aged ≥ 19 years, relapsed or refractory patients treated with ibrutinib, including relapse after autologous stem cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival period | Up to 3 years, From the date of diagnosis with MCL to the date of relapse/disease progression, or last follow-up date
  Progression free survival period with ibrutinib

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years, From the date of diagnosis with MCL to the date of death, or last follow-up date
  Overall response rate with ibrutinib

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, Professor, Principal Investigator — Samsung Medical Center
Locations (1):
- 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided